CLINICAL TRIAL: NCT00789854
Title: A Randomised, 6-week, Multicentre, Open-label, Rater-blinded Parallel Group Study Comparing Quetiapine Extended Release Monotherapy and Augmentation With Lithium Augmentation in Patients With Treatment Resistant Depression
Brief Title: Comparing Quetiapine XR Monotherapy and Augmentation With Lithium Augmentation in TRD Patients
Acronym: RUBY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00044
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-04

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
Keywords: Depression; MDD; TRD
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression | interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Add-on Quetiapine XR+SSRI/Venlafaxine (Active Comparator): Selective serotonin reuptake inhibitors (SSRI) or Venlafaxine from previous therapy + add-on treatment with quetiapine XR, 300mg tablet once daily (od).
  From previous anti-depressant treatment 64% of the patients had SSRI and 35% had Venlafaxine at baseline.
  Interventions: Drug: Quetiapine XR; Drug: SSRI/Venlafaxine
- Add-on Lithium+SSRI/Venlafaxine (Active Comparator): Selective serotonin reuptake inhibitors (SSRI) or venlafaxine from previous therapy + add-on treatment with lithium, approximately 900mg tablet once daily (od).
  From previous anti-depressant treatment 67% of the patients had SSRI and 33% had Venlafaxine at baseline.
  Interventions: Drug: Lithium carbonate; Drug: SSRI/Venlafaxine
- Monotherapy Quetiapine XR (Active Comparator): Switch from previous treatment with SSRI or venlafaxine to quetiapine XR monotherapy, 300mg tablet once daily (od)
  Interventions: Drug: Quetiapine XR

INTERVENTIONS:
Drug: Quetiapine XR — 300 mg once daily (od)
  Other Names: Seroquel XR
  Arms: Add-on Quetiapine XR+SSRI/Venlafaxine; Monotherapy Quetiapine XR
Drug: Lithium carbonate — 900 mg once daily (od)
  Other Names: Quilonum Retard
  Arms: Add-on Lithium+SSRI/Venlafaxine
Drug: SSRI/Venlafaxine — SSRI - doses within label, Venlafaxine dose up to 225 mg/day
  Arms: Add-on Lithium+SSRI/Venlafaxine; Add-on Quetiapine XR+SSRI/Venlafaxine

SUMMARY:
The primary objective of the study is to evaluate the efficacy of Quetiapine extended release (XR) in combination with an selective serotonin reuptake inhibitor (SSRI) or Venlafaxine versus Lithium in combination with an selective serotonin reuptake inhibitor or Venlafaxine versus Quetiapine extended release monotherapy in subjects with treatment resistant depression as assessed by the changes from randomisation to week 6 in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score. As an independent objective, the primary objective will also be evaluated in two subgroups of patients: (1) patients who were resistant to two previous antidepressant therapies and (2) in the subgroup of patients with one previous failure.

DETAILED DESCRIPTION:
The secondary objectives of the study are to compare the effects of the three different treatment regimen as assessed by the following variables and, if applicable, by their changes from randomisation to week 6 (end of study). Additionally the time of onset of therapeutic effect will be assessed by evaluating efficacy data after the first four days (Day 4) of treatment as well as after the first week of treatment (Day 8). These analyses will also be performed in the subgroups of patients with 2 failed previous antidepressants and patients with 1 failure.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical diagnosis as confirmed by the M.I.N.I. meeting criteria from the Diagnostic and Statistical Manual of Mental disorders, 4th Edition (DSM-IV) for any of the following:296.2x MDD, Single Episode296.3x MDD, Recurrent Episode
* Current episode of depression present, at least 42 days prior to enrolment but not more than 18 months
* MADRS-Score ≥ 25 at enrolment and randomisation

Exclusion Criteria:

* Patients with a DSM-IV Axis I disorder other than MDD within 6 months of randomisation
* Patients with a diagnosis of DSM-IV Axis II disorder which has a major impact on the patient's current psychiatric status
* Patients who, in the investigator's judgment pose a current serious suicidal or homicidal risk, or have made a suicide attempt within the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bauer, professor, Principal Investigator — Germany; Birgit Ekholm, PhD, Study Director — AstraZeneca MC Sweden
Locations (106):
- Australia (11):
  - Research Site, Garran, Australian Capital Territory
  - Research Site, Brisbane, Queensland
  - Research Site, Everton Park, Queensland
  - Research Site, Townsville, Queensland
  - Research Site, Gilberton, South Australia
  - Research Site, Clayton, Victoria
  - Research Site, Frankston, Victoria
  - Research Site, Heidelberg, Victoria
  - Research Site, Malvern, Victoria
  - Research Site, Prahran, Victoria
  - Research Site, Richmond, Victoria
- Austria (6):
  - Research Site, Graz
  - Research Site, Klagenfurt
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Wels
  - Research Site, Wiener Neustadt
- Belgium (4):
  - Research Site, Assebroek, Belgium
  - Research Site, Diest, Belgium
  - Research Site, Liège, Belgium
  - Research Site, Tielt
- Bulgaria (7):
  - Research Site, Cerova Koria Village, Veliko Tarnovo
  - Research Site, Kardzhali
  - Research Site, Pazardzhik
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Denmark (3):
  - Research Site, Esbjerg N
  - Research Site, Frederiksberg
  - Research Site, Odense
- Germany (32):
  - Research Site, Aachen
  - Research Site, Achim
  - Research Site, Augsburg
  - Research Site, Bad Homburg
  - Research Site, Bad Honnef
  - Research Site, Bad Saarow
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Bochum
  - Research Site, Butzbach
  - Research Site, Chemnitz
  - Research Site, Dresden
  - Research Site, Düren
  - Research Site, Düsseldorf
  - Research Site, Ellwangen
  - Research Site, Erbach im Odenwald
  - Research Site, Gelsenkirchen
  - Research Site, Gütersloh
  - Research Site, Halle
  - Research Site, Hattingen
  - Research Site, Herborn
  - Research Site, Kassel
  - Research Site, Köthen
  - Research Site, Neu-Isenburg
  - Research Site, Neubrandenburg
  - Research Site, Nuremberg
  - Research Site, Oldenburg
  - Research Site, Ostfildern
  - Research Site, Schwerin
  - Research Site, Stuttgart
  - Research Site, Westerstede
  - Research Site, Würzburg
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Nyíregyháza
- Italy (9):
  - Research Site, Brixen, BZ
  - Research Site, Bruneck, BZ
  - Research Site, Cagliari, CA
  - Research Site, Pisa, PI
  - Research Site, Roma, RM
  - Research Site, Bolzano
  - Research Site, Catania
  - Research Site, Napoli
  - Research Site, Roma
- Portugal (4):
  - Research Site, Braga
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Santarém
- Romania (4):
  - Research Site, Galati, Galați County
  - Research Site, Bucharest
  - Research Site, Craiova
  - Research Site, Sibiu
- Slovakia (9):
  - Research Site, Bratislava
  - Research Site, Krupina
  - Research Site, Levice
  - Research Site, Liptovský Mikuláš
  - Research Site, Michalovce Stranany
  - Research Site, Prešov
  - Research Site, Rožňava
  - Research Site, Zilina-bytcica
  - Research Site, Zlaté Moravce
- Spain (5):
  - Research Site, Salamanca, Castille and León
  - Research Site, Zamora, Castille and León
  - Research Site, Barcelona, Catalonia
  - Research Site, Vigo, Galicia
  - Research Site, Langreo, Principality of Asturias
- United Kingdom (8):
  - Research Site, Addlestone, Surrey
  - Research Site, Winnick, Warrington
  - Research Site, Horsham, West Sussex
  - Research Site, Coventry
  - Research Site, Glasgow
  - Research Site, Harrow
  - Research Site, Hull
  - Research Site, Winsford

REFERENCES:
- [Derived] Bauer M, Dell'osso L, Kasper S, Pitchot W, Dencker Vansvik E, Kohler J, Jorgensen L, Montgomery SA. Extended-release quetiapine fumarate (quetiapine XR) monotherapy and quetiapine XR or lithium as add-on to antidepressants in patients with treatment-resistant major depressive disorder. J Affect Disord. 2013 Oct;151(1):209-19. doi: 10.1016/j.jad.2013.05.079. Epub 2013 Jun 27. PMID 23810357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 3 arm, open-label randomised, rater blinded, parallel group study comparing quetiapine XR monotherapy and augmentation with lithium augmentation in patients with treatment resistant depression, Recruitment period 6 November 2008 to 19 June 2009
Pre-assignment Details: At visit 1 and 2 (randomisation) the patients should have a Montgomery-Asberg Depression Rating Scale (MADRS) total score above or equal to 25
Groups:
- Quetiapine XR Mono: Switch from previous treatment with SSRI or venlafaxine to quetiapine XR monotherapy, 300mg tablet once daily (od)
- Add-on Quetiapine XR: Selective serotonin reuptake inhibitors (SSRI) or venlafaxine from previous therapy + add-on treatment with quetiapine XR, 300mg tablet once daily (od)
- Add-on Lithium: Selective serotonin reuptake inhibitors (SSRI) or venlafaxine from previous therapy + add-on treatment with lithium, approximately 900mg tablet once daily (od)
Period: Overall Study
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Started | 228 | 231 | 229
Completed | 179 | 196 | 182
Not Completed | 49 | 35 | 47
Not completed — Adverse Event | 28 | 23 | 18
Not completed — Lost to Follow-up | 1 | 1 | 4
Not completed — Withdrawal by Subject | 9 | 6 | 17
Not completed — Eligibility criteria not fulfilled | 2 | 5 | 1
Not completed — Severe non-compliance to the protocol | 3 | 0 | 0
Not completed — Safety reasons | 0 | 0 | 2
Not completed — Other | 6 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium | Total
Number analyzed (Participants) | 225 | 229 | 221 | 675
Age Continuous [Mean (Full Range); unit: years] — Baseline characteristics are presented using the ITT population (Quetiapine XR mono 225 participants, Add-on Quetiapine XR 229 participants and Add-on Lithium 221 participants) and not all randomized patients
  years | 47 [20 to 65] | 47 [20 to 67] | 47 [19 to 67] | 47 [19 to 67]
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics are presented using the ITT population (Quetiapine XR mono 225 participants, Add-on Quetiapine XR 229 participants and Add-on Lithium 221 participants) and not all randomized patients
  Participants
    Female | 152 | 162 | 152 | 466
    Male | 73 | 67 | 69 | 209
Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) [Number; unit: Participants]
  Diagnose code 296.2x Major Depressive Disorder (MD | 50 | 36 | 41 | 127
  Diagnose code 296.3x MDD, Recurrent | 175 | 193 | 180 | 548
Montgomery-Asberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: Units on a scale] — Units on a scale from 0 to 60. Lower score indicates a better health status.
  Units on a scale | 33.74 (5.6) | 33.15 (5.34) | 32.91 (5.2) | 33.32 (5.4)
Weight [Mean (Standard Deviation); unit: kg] | 75.3 (17.2) | 75.2 (17) | 76.4 (16.1) | 75.8 (16.65)

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressive Symptoms Between Randomisation and Week 6 Measured by Change in Montgomery Asberg Depression Rating Scale (MADRS) Total Score (Per Protocol Analysis Set)
Description: Change in LS mean total Montgomery Asberg Depression Rating Scale (MADRS) score from randomisation to end-of-treatment (week 6) (Scale 0-60), lower score indicates a better health status.
Time Frame: 6 weeks treatment
Population: Analysis was 'per protocol'. Exclusion reason from analysis: Violation of exclusion/inclusion criteria; Non-compliance regarding prohibited concomitant medication, Total unavailability of MADRS score after randomization, Patient not treated with any dose of study drug after randomization, Non-compliance regarding titration to 300 mg quetiapine/d.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 180 | 183 | 109
scores on a scale | -16.2 (0.843) [lower limit 0.843] | -17.2 (0.826) [lower limit 0.826] | -14.9 (0.97) [lower limit 0.97]
Statistical Analysis 1: Comparison: Add-on Quetiapine XR vs Add-on Lithium; Add-on quetiapine XR was tested versus add-on lithium for non-inferiority. The null hypothesis was that the add-on quetiapine treatment was non-inferior to add-on lithium; Test type: Non-Inferiority or Equivalence — The non-inferiority margin for differences was set to 3 units in the MADRS total score. A power set to 80% and using a Bonferroni-adjusted one-sided alpha* = alpha/3 = 0.0083 yields a planned sample size of 192 patients per study group. With a drop out of 4% a total of 600 randomized patients were required to obtain 192 efficacy evaluable patients per treatment group; ANCOVA — The CI is for comparing add-on quetiapine versus add-on Lithium. The CI = confidence interval was adjusted for multiple comparisons. The -0.05 value should have been +3 or above to fail to reject the null hypothesis; Non-inferiority between add-on quetiapine XR and add-on lithium was shown in the Per Protocol analysis set; Mean Difference (Final Values) = -2.322, 97.5% CI [-4.6 to -0.05]
Statistical Analysis 2: Comparison: Quetiapine XR Mono vs Add-on Lithium; Quetiapine XR mono was tested versus add-on lithium for non-inferiority. The null hypothesis was that the quetiapine XR mono treatment was non-inferior to add-on lithium; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA — The CI is for comparing quetiapine XR mono versus add-on Lithium. The CI = confidence interval was adjusted for multiple comparisons. The 1.312 value should have been +3 or above to fail to reject the null hypothesis; Non-inferiority between quetiapine XR mono and add-on lithium was shown in the Per Protocol analysis set; Mean Difference (Final Values) = -1.639, 97.5% CI [-3.24 to 1.312]

2. Primary Outcome: Change in Depressive Symptoms Between Randomisation and Week 6 Measured by Change in Montgomery Asberg Depression Rating Scale (MADRS) Total Score (Modified Intention to Treat Analysis Set)
Description: as for outcome 1
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 225 | 229 | 221
scores on a scale | -13.9 (0.806) [lower limit 0.806] | -15.1 (0.797) [lower limit 0.797] | -13.3 (0.801) [lower limit 0.801]
Statistical Analysis 1: Comparison: Add-on Quetiapine XR vs Add-on Lithium; The null hypothesis was that the add-on quetiapine XR treatment was not different to the add-on lithium treatment. The power calculation was done for the primary non-inferior analysis. This superiority analysis was only done if the non-inferior analysis was successful; Test type: Superiority or Other; p = 0.0489, ANCOVA — Adjustment for multiplicity was done, alpha = 0.025; Superiority testing of primary outcome showed no significant difference in the Modified Intention To Treat (ITT) population
Statistical Analysis 2: Comparison: Quetiapine XR Mono vs Add-on Lithium; The null hypothesis was that the quetiapine XR mono treatment was not different from the add-on lithium treatment. The power calculation was done for the primary non-inferior analysis. This superiority analysis was only done if the non-inferior analysis was successful; Test type: Superiority or Other; p = 0.4368, ANCOVA — Adjustment for multiplicity was done, alpha = 0.025; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Depression Remission; Montgomery-Asberg Depression Rating Scale MADRS ≤10, All Patients
Description: Number of patients in remission, with total Montgomery Asberg Depression Rating Scale (MADRS) score ≤10. MADRS scale has range from 0 to 60, where the lower score indicates the better health status.
Time Frame: 6 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 225 | 229 | 221
Participants | 53 | 73 | 60

4. Secondary Outcome: Depression Remission; Montgomery-Asberg Depression Rating Scale (MADRS) ≤10, Patients With One Previous Treatment Failure
Description: Number of patients in remission with one previous treatment failure and with total Montgomery Asberg Depression Rating Scale (MADRS) score ≤10. MADRS scale has range from 0 to 60, where the lower score indicates the better health status.
Time Frame: 6 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 114 | 117 | 114
Participants | 22 | 42 | 31

5. Secondary Outcome: Depression Remission; Montgomery-Asberg Depression Rating Scale (MADRS) ≤10, Patients With Two Previous Treatment Failure
Description: Number of patients in remission with two previous treatment failure and with total Montgomery Asberg Depression Rating Scale (MADRS) score ≤10. MADRS scale has range from 0 to 60, where the lower score indicates the better health status.
Time Frame: 6 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 114 | 114 | 115
Participants | 31 | 31 | 29

6. Secondary Outcome: Depression Remission; Montgomery-Asberg Depression Rating Scale (MADRS) ≤8
Description: Number of patients in remission with total Montgomery Asberg Depression Rating Scale (MADRS) score ≤8. MADRS scale has range from 0 to 60, where the lower score indicates the better health status.
Time Frame: 6 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 225 | 229 | 221
Participants | 35 | 58 | 45

7. Secondary Outcome: Depression Remission; Montgomery-Asberg Depression Rating Scale (MADRS) ≤12
Description: Number of patients in remission with total Montgomery Asberg Depression Rating Scale (MADRS) score ≤12. MADRS scale has range from 0 to 60, where the lower score indicates the better health status.
Time Frame: 6 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 225 | 229 | 221
Participants | 67 | 89 | 73

8. Secondary Outcome: Response Rate; Montgomery-Asberg Depression Rating Scale (MADRS) Score Reduced ≥ 50%, All Patients
Description: Response rate at end of study measured as number of patients with Montgomery Asberg Depression Rating Scale (MADRS) with total score reduction ≥ 50% compared to baseline, the higher number of patients the better
Time Frame: 6 week of treatments
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 225 | 229 | 221
Participants | 114 | 120 | 102

9. Secondary Outcome: Response Rate; Montgomery-Asberg Depression Rating Scale (MADRS) Score Reduced ≥ 50%, Patients With One Previous Treatment Failure
Description: as for outcome 8
Time Frame: 6 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 114 | 117 | 114
Participants | 54 | 65 | 53

10. Secondary Outcome: Response Rate; Montgomery-Asberg Depression Rating Scale (MADRS) Score Reduced ≥ 50%, Patients With Two Previous Treatment Failure
Description: as for outcome 8
Time Frame: 6 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 114 | 114 | 115
Participants | 60 | 55 | 49

11. Secondary Outcome: Responder: Clinical Global Impression Improvement (CGI-I) Item 2, All Patients
Description: Change in global improvement measured by Clinical Global Impression Improvement (CGI-I). Scale from 1-4, where lower value shows a larger improvement.
Time Frame: 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 224 | 229 | 220
scores on a scale | -1.54 (1.24) | -1.85 (1.34) | -1.58 (1.32)

12. Secondary Outcome: Responder: Clinical Global Impression Improvement (CGI)-I Item 2, Patients With One Previous Treatment Failure
Description: Change in global improvement measured by Clinical Global Impression Improvement (CGI-I). Scale from 1-4, where a lower value shows a larger improvement.
Time Frame: 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 113 | 115 | 111
scores on a scale | -1.42 (1.17) | -1.91 (1.31) | -1.62 (1.27)

13. Secondary Outcome: Responder: Clinical Global Impression Improvement (CGI-I) Item 2, Patients With Two Previous Treatment Failure
Description: as for outcome 12
Time Frame: 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 111 | 114 | 109
scores on a scale | -1.67 (1.30) | -1.79 (1.36) | -1.54 (1.38)

14. Secondary Outcome: Change in Clinical Global Impression Scale (CGI-S), All Patients
Description: Change in severity of illness measured by Clinical Global Impression Scale (CGI-S). Scale form 1-7, where a lower value shows a larger improvement.
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 224 | 229 | 220
scores on a scale | -1.43 (0.101) [lower limit 0.101] | -1.65 (0.099) [lower limit 0.099] | -1.49 (0.1) [lower limit 0.1]

15. Secondary Outcome: Change in Clinical Global Impression Scale (CGI-S), Patients With One Previous Treatment Failure
Description: Change in severity of illness measured by Clinical Global Impression Scale (CGI-S). Scale from 1-7, where a lower value shows a larger improvement.
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 113 | 115 | 111
scores on a scale | -1.45 (0.133) [lower limit 0.133] | -1.82 (0.13) [lower limit 0.13] | -1.59 (0.13) [lower limit 0.13]

16. Secondary Outcome: Change in Clinical Global Impression Scale (CGI-S), Patients With Two Previous Treatment Failure
Description: as for outcome 15
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 111 | 114 | 109
scores on a scale | -1.52 (0.133) [lower limit 0.133] | -1.55 (0.131) [lower limit 0.131] | -1.45 (0.135) [lower limit 0.135]

17. Secondary Outcome: Change in Beck Depression Inventory (BDI)
Description: Self-rating assessment of depressive symptoms using Beck Depression Inventory (BDI). Scale from 0-63, where a lower value shows a larger improvement.
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 213 | 212 | 205
scores on a scale | -11.7 (0.926) [lower limit 0.926] | -13.5 (0.921) [lower limit 0.921] | -12.2 (0.922) [lower limit 0.922]

18. Secondary Outcome: Change in Pain, Measured by Visual Analog Scale (VAS)
Description: Self-rating assessment of pain using a visual analogue scale (VAS). Scale from 0-100, where a lower value shows a larger improvement.
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 221 | 222 | 218
scores on a scale | -9.47 (1.695) [lower limit 1.695] | -8.03 (1.681) [lower limit 1.681] | -8.3 (1.682) [lower limit 1.682]

19. Secondary Outcome: Change in Anxiety Measured by Visual Analog Scale (VAS)
Description: Self-rating assessment of anxiety using a visual analogue scale (VAS). Scale from 0-100, where a lower value shows a larger improvement.
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 219 | 224 | 218
scores on a scale | -21.2 (1.972) [lower limit 1.972] | -23.4 (1.947) [lower limit 1.947] | -20.6 (1.952) [lower limit 1.952]

20. Secondary Outcome: Change in Anxiety Measured by State-Trait Anxiety Inventory (STAI), State Anxiety Inventory
Description: Self-rating assessment of anxiety measured by STAI, state anxiety inventory (Scale 20-80, where a lower value shows a larger improvement)
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 223 | 227 | 217
Scores on a scale | -0.62 (0.347) [lower limit 0.347] | 0.014 (0.344) [lower limit 0.344] | -0.87 (0.35) [lower limit 0.35]

21. Secondary Outcome: Change in Anxiety Measured by STAI, Trait Anxiety Inventory
Description: Self-rating assessment of anxiety measured by State-Trait Anxiety Inventory (STAI), trait anxiety inventory (Scale 20-80, where a lower value shows a larger improvement)
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 220 | 220 | 214
Scores on a scale | -1.01 (0.331) [lower limit 0.331] | -1.36 (0.328) [lower limit 0.328] | -1.39 (0.331) [lower limit 0.331]

22. Secondary Outcome: Change in Sleep Quality Measured by Montgomery Asberg Depression Rating Scale (MADRS), Item 4
Description: Sleeping quality measured by Montgomery-Asberg Depression Rating Scale (MADRS) item 4 (reduced sleep) (Scale 0-6, where a lower value shows a larger improvement)
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: MADRS item 4 score
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 225 | 229 | 221
MADRS item 4 score | -2.2 (0.108) [lower limit 0.108] | -2.4 (0.107) [lower limit 0.107] | -1.63 (0.108) [lower limit 0.108]

23. Secondary Outcome: Change in Sleep Quality Measured by Pittsburgh Sleep Quality Index (PSQI)
Description: Self-rated sleeping quality measured by PSQI (Scale 0-21, subscales 0-3, 18 questions, where a lower value shows a larger improvement)
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 200 | 196 | 185
Scores on a scale | -4.77 (0.36) [lower limit 0.36] | -4.96 (0.358) [lower limit 0.358] | -3.51 (0.364) [lower limit 0.364]

24. Secondary Outcome: Change in Quality of Life Measured by Short-form Health Survey (SF-36), Mental Component
Description: Self rating assessment of quality in life using SF-36, mental component (Scale 0-100, where a higher value shows a larger improvement)
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 178 | 171 | 174
Scores on a scale | 9.59 (0.929) [lower limit 0.929] | 10.77 (0.925) [lower limit 0.925] | 9.66 (0.932) [lower limit 0.932]

25. Secondary Outcome: Change in Quality of Life Measured by Short-form Health Survey (SF-36), Physical Component
Description: Self rating assessment of quality in life using SF-36, physical component (Scale 0-100, where a higher value shows a larger improvement)
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 178 | 171 | 174
Scores on a scale | 5.224 (0.811) [lower limit 0.811] | 5.065 (0.813) [lower limit 0.813] | 4.566 (0.817) [lower limit 0.817]

26. Secondary Outcome: Change in Quality of Life Measured by Health Questionnaire EQ-5D as Utility
Description: Self rating assessment of quality in life using EQ-5D utility (Scale 0-100, where a higher value shows a larger improvement)
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 220 | 220 | 215
Scores on a scale | 0.184 (0.023) [lower limit 0.023] | 0.224 (0.023) [lower limit 0.023] | 0.208 (0.023) [lower limit 0.023]

27. Secondary Outcome: Change in Work Productivity and Activity Impairment: General Health (WPAI:GH)
Description: Self rating assessment of working productivity using WPAI:GH (Scale 0 to number of hours worked during a week multiplied with the salary in Euro, a lower value shows a larger improvement)
Time Frame: 6 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 31 | 39 | 25
Scores on a scale | -233 (0.023) [lower limit 79.09] | -185 (0.023) [lower limit 72.38] | -299 (0.023) [lower limit 87.42]

28. Secondary Outcome: Change in Clinical Global Impression (CGI) Item 4 Efficacy and Safety Combined, All Patients
Description: The physician has evaluated the therapeutic effect and the side effect combined at end of study. Patients with a 'marked/moderate' therapeutic effect and 'None/Do Not Significantly Interfere' side effect has been added. The higher values show more patients with a treatment effect without any side-effect. The range is from 0 patients to the maximum number of patients in the treatment arm (225, 229 or 221).
Time Frame: 6 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 225 | 229 | 221
Participants | 135 | 146 | 131

29. Secondary Outcome: Change in Clinical Global Impression (CGI) Item 4 Efficacy and Safety Combined, Patients With One Previous Treatment Failure
Description: The physician has evaluated the therapeutic effect and the side effect combined at end of study. Patients with a 'marked/moderate' therapeutic effect and 'None/Do Not Significantly Interfere' side effect has been added. The higher values show more patients with a treatment effect without any side-effect. The range is from 0 patients to the maximum number of patients in the treatment arm.
Time Frame: 6 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 113 | 115 | 111
Participants | 67 | 75 | 69

30. Secondary Outcome: Change in Clinical Global Impression (CGI) Item 4 Efficacy and Safety Combined, Patients With Two Previous Treatment Failures
Description: as for outcome 29
Time Frame: 6 week of treatments
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Number analyzed (Participants) | 112 | 114 | 110
Participants | 68 | 71 | 62

ADVERSE EVENTS:
Arm/Group | Quetiapine XR Mono | Add-on Quetiapine XR | Add-on Lithium
Serious Adverse Events (participants affected / at risk) | 5/228 | 5/231 | 2/229
Other Adverse Events (participants affected / at risk) | 93/228 | 90/231 | 41/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR Mono (N=228) | Add-on Quetiapine XR (N=231) | Add-on Lithium (N=229)
Depression (Psychiatric disorders) | 0 | 3 | 1
Affective Disorder (Psychiatric disorders) | 1 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Mania (Psychiatric disorders) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR Mono (N=228) | Add-on Quetiapine XR (N=231) | Add-on Lithium (N=229)
Somnolence (Nervous system disorders) | 22 | 20 | 0
Sedation (Nervous system disorders) | 15 | 11 | 0
Tremor (Nervous system disorders) | 0 | 0 | 15
Dizziness (Nervous system disorders) | 11 | 14 | 0
Headache (Nervous system disorders) | 11 | 10 | 13
Fatigue (General disorders) | 21 | 13 | 7
Dry mouth (Gastrointestinal disorders) | 13 | 22 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less